CLINICAL TRIAL: NCT00835744
Title: Among Non-IVF Patients Undergoing Ovulation Induction With Clomiphene Citrate (Clomid® 50 mg), Does Administration of an Increased Dose of Clomiphene Citrate (Clomid® 100 mg) Compared With Gonadotropins, Achieve Similar Rates of Folliculogenesis?
Brief Title: Comparison of Clomiphene Citrate and Gonadotropins in Ovulation Induction Cycles
Acronym: cc versus FSH
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Principal Investigator, Blockeel Christophe, Dr, Universitair Ziekenhuis Brussel
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2008/192
Record Dates: First submitted 2009-02-03; First posted 2009-02-04 (Estimated); Last update posted 2012-03-28 (Estimated); Status verified 2012-03

CONDITIONS: Infertility
Keywords: ovulation induction; clomiphene citrate; gonadotropins
MeSH Terms: conditions — Infertility | interventions — Clomiphene; Gonadotropins

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Placebo Comparator): Patients undergo a standard treatment with clomiphene citrate from day 3 until day 7 of the cycle at a dose of 50 mg daily. If no reaction on day 13 of the cycle, an increased dose of 100 mg of clomiphene citrate is administered from day 13 until day 17 of the cycle.
  Interventions: Drug: clomiphene citrate
- B (Active Comparator): Patients undergo a standard treatment with clomiphene citrate from day 3 until day 7 of the cycle at a dose of 50 mg daily. If no reaction on day 13 of the cycle, gonadotropins (75IU) are administered from day 13 until day 17 of the cycle.
  Interventions: Drug: gonadotropins

INTERVENTIONS:
Drug: clomiphene citrate — ovulation induction
  Arms: A
Drug: gonadotropins — ovulation induction
  Arms: B

SUMMARY:
The purpose of the present study is to analyse prospectively if highly purified hMG compared with increased dose of clomiphene citrate has different outcomes in folliculogenesis in ovulation induction cycles.

ELIGIBILITY:
Inclusion Criteria:

* < 39 years old on day of randomisation
* FSH < 12 (in the early follicular phase)
* Normal ultrasound scan, i.e. presence of both ovaries, without evidence of abnormality within 6 months prior to randomisation.
* Chronic oligo or anovulation (WHO 2)
* BMI between 18 and 31 (both inclusive)

Exclusion Criteria:

* ≥ 39 years old on day of randomisation

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2008-08; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
folliculogenesis | april 2009

SECONDARY OUTCOMES:
pregnancy rate | april 2009

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Brussel, Jette, Belgium